CLINICAL TRIAL: NCT05173480
Title: Does Virtual Reality Rehabilitation Added to Conventional Physiotherapy Improve Mobility, Balance, and Walking Assessed by Timed Up and Go in Patients With Total Hip Arthroplasty? A Randomized Controlled Trial
Brief Title: Does Virtual Reality Rehabilitation Improve Mobility, Balance, and Walking in Patients With Total Hip Arthroplasty?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mauro Crestani (Other Government)
Responsible Party: Sponsor-Investigator, Mauro Crestani, Principal Investigator, Azienda Ulss 9 Scaligera
Organization: Azienda Ulss 9 Scaligera (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AziendaU9S
Record Dates: First submitted 2021-12-08; First posted 2021-12-30 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Total Hip Arthroplasty
Keywords: Virtual reality rehabilitation; Physiotherapy; Physical therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): VRRS rehabilitation exercise therapy through a virtual reality rehabilitation system in addition to conventional rehabilitation.
  Interventions: Other: Conventional rehabilitation; Device: Virtual Reality Rehabilitation System (VRRS)
- Control group (Active Comparator): VRRS rehabilitation exercise therapy through a virtual reality rehabilitation system, with sensors not connected, in addition to conventional rehabilitation.
  Interventions: Other: Conventional rehabilitation; Device: Virtual Reality Rehabilitation System (VRRS)

INTERVENTIONS:
Other: Conventional rehabilitation — Exercise therapy through conventional rehabilitation training made by physiotherapists.
Device: Virtual Reality Rehabilitation System (VRRS) — Exercise therapy through a virtual reality rehabilitation system (VRRS).
  Arms: Experimental group
Device: Virtual Reality Rehabilitation System (VRRS) — Exercise therapy through a virtual reality rehabilitation system (VRRS) with sensors not connected.
  Arms: Control group

SUMMARY:
This study aims to assess the efficacy of virtual reality through the Virtual Reality Rehabilitation System (VRRS) added to conventional rehabilitation versus conventional rehabilitation alone, for improving mobility, balance, and walking assessed by Timed Up and Go after primary Total Hip Arthroplasty.

DETAILED DESCRIPTION:
Following ethics approval by the ULSS 9, adults with THA (at 7 days after surgery), aged between 45 and 85 years old will be recruited for the study by the office worker of the rehabilitation hospital. Patients will be informed about the aim of the study and will sign the informed consent. Patients that decided to participate in the study will be randomized into two rehabilitation groups: experimental group and control group. Patients will be evaluated for reaching the baseline data from a physiotherapist blind to the aim of the study. Both groups (experimental and control) will receive the same clinical indications during hospitalization. Both groups will perform the same daily warm-up exercises supervised by physiotherapists external to the study investigation and will receive the same conventional-exercises program. In addition to this, each group will perform a second rehabilitation session with the virtual reality, using the Virtual Reality Rehabilitation System (VRRS), but in the control group, the sensors of VRRS will be not connected. The primary outcome will be the Timed Up and Go (TUG), the test used to assess mobility, balance, and walking.

ELIGIBILITY:
Inclusion Criteria:

* age: 45-85 years
* primary unilateral THA for hip osteoarthritis
* signed informed consent

Exclusion Criteria:

* people with clinically unstable serious diseases (e.g., heart or lung disease)
* secondary THA replacement on the same side
* hip replacement for neoplasm, proximal femoral fracture, or other causes out of osteoarthritis
* contemporary bilateral replacement
* cancer
* presence of neurological diseases previous or following surgery
* congenital abnormalities
* patients with THA infection
* diabetes
* psychotropic drugs assumption for pain management

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Timed Up and Go (TUG) score | baseline (7 days after surgery) and at discharge (28 days after surgery)
  The TUG is a timed test used to assess mobility, balance, and walking. The subject must stand up from a chair, walk a distance of 3 meters, turn around, walk back to the chair and sit down - all performed as quickly and as safely as possible.

SECONDARY OUTCOMES:
Change in the Hip dysfunction and Osteoarthritis Outcome Score (HOOS) | baseline (7 days after the surgery), at discharge (28 days after surgery) and at 6 months after surgery (by telephone interview)
  The HOOS scale scores range from 0 to 100 (0: total hip disability, 100: perfect hip health)
Change in the Numeric Rating Scale for pain (NPRS) | baseline (7 days after surgery), at discharge (28 days after surgery) and at 6 months
  A 10-cm Numerical Pain Rating Scale (0: no pain, 10: maximum pain) will be used to assess the current level of hip pain before rehabilitation treatment.
Change in the Hip Active Range of Motion | baseline (7 days after surgery) and at discharge (28 days after surgery)
  Assessed by goniometer (degree of movement)
Change in the Strength of main muscles of the pelvis and thigh of the affected limb | baseline (7 days after surgery) and at discharge (28 days after surgery)
  Assessed by dynamometer
Change in the 6 Minutes Walking Test (6MWT) | baseline (7 days after surgery) and at discharge (28 days after surgery)
  Walking ability and cardio-respiratory function
Change in the Short Form Health Survey 36 (SF-36) | baseline (7 days after surgery) and at discharge (28 days after surgery) and at 6 months (telephone interview)
  Short Form Health Survey scores range from 0 to 100 (0: maximum disability; 100: no disability)
Change in the Numeric Rating of Patient Satisfaction with functional outcome | assessed and reported at discharge (28 days after surgery) at 6 months (telephone interview)
  A 10-cm Numeric Rating of Patient Satisfaction with the functional outcome (0: no satisfaction; 10: maximum satisfaction) is used to assess the general satisfaction of the patients
The drugs assumption for pain management | assessed and reported at discharge (28 days after surgery)
  Type of drugs intake for each group during rehabilitation recovery

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Crestani, Principal Investigator — Azienda Ulss 9 Scaligera
Locations (1):
- AULSS 9 - Marzana Hospital, Verona, Italy